CLINICAL TRIAL: NCT05582850
Title: A Phase 1, Multicentre, Open-label, Dose-escalation and Expansion Study to Determine a Recommended Phase 2 Dose (RP2D) of DT-9081 in Participants With Advanced Solid Tumours
Brief Title: DT-9081 Study in Participants With Advanced, Recurrent or Metastatic Solid Tumours
Acronym: EPRAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Domain Therapeutics SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DT-9081-CLI-001
Record Dates: First submitted 2022-10-10; First posted 2022-10-17 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Solid Tumor, Adult
Keywords: Advanced cancer; Immuno-oncology

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DT-9081 (Experimental): Capsule, 25 mg, 50 mg and 100 mg
  Interventions: Drug: DT-9081 - dose escalation; Drug: DT-9081 - expansion

INTERVENTIONS:
Drug: DT-9081 - dose escalation — Patients will be dosed orally once daily. The schedule might be adjusted in case of toxicities.
  Other Names: Phase 1 dose-escalation part
Drug: DT-9081 - expansion — A homogeneous patient population will receive DT-9081 at up to 3 dose levels.
  Other Names: Phase 1 expansion part

SUMMARY:
This is a Phase 1, multicentre, open-label, dose-escalation study to determine a recommended phase 2 dose (RP2D) of DT-9081, followed by an expansion study of DT-9081 in participants with advanced, recurrent or metastatic solid tumours

DETAILED DESCRIPTION:
This first-in-human Phase 1, multicentre, open label study is evaluating the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary efficacy of DT-9081 in adult patients with advanced, recurrent or metastatic solid tumours who failed standard of care therapies.

This Phase 1 study consists of 2 parts. The first part is a dose-escalation using a modified 3+3 design with up to 8 dose escalation cohorts at increasing levels. The dose-escalation part aims at determining the recommended phase 2 dose. The second part is an expansion to validate the dose/schedule of administration as well as to assess preliminary efficacy of DT-9081.

Patients will be dosed orally once daily. The schedule might be adjusted in case of toxicities.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a histologically or cytologically confirmed advanced solid tumour that is locally advanced (i.e., not eligible for curative surgery or radiotherapy), recurrent or metastatic, and who have failed or are ineligible for standard of care therapies.
* Participants must be ≥18 years of age.
* Participants must have measurable disease per RECIST v1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* Participants must have adequate organ function.

Exclusion Criteria:

* Participants using drugs interfering with the COX-2 pathways or prohibited drugs.
* Participants with unresolved AEs from previous anti-cancer therapies of Grade ≥ 2 with exception of alopecia. Participants with Grade ≤ 2 neuropathy may be eligible.
* Participants who underwent major surgery or significant traumatic injury within 4 weeks prior to Cycle 1 Day 1 who have not recovered adequately from any AEs and/or complications from the intervention prior to starting study drug.
* Participants who have received prior radiotherapy within the last 4 weeks before start of study drug treatment (limited field palliative radiotherapy within 2 weeks).
* Participants who have already received EP4R antagonist in an investigational trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2022-11-24 (Actual); Primary Completion 2025-04-08 (Actual); Study Completion 2025-07-28 (Actual)

PRIMARY OUTCOMES:
Dose escalation: recommended phase 2 dose (RP2D) | Cycle 1 (28 days)
  The RP2D of DT-9081 is determined using pharmacokinetics, pharmacodynamics and safety data of the dose escalation part of the study.
Dose escalation: safety assessment | Cycle 1 (28 days)
  Number of dose-limiting toxicities (DLTs).
Dose escalation and expansion: safety assessment | From the first dose of study drug up to 30 days after the last dose of study drug
  Incidence and severity of treatment-emergent AEs (TEAEs) and treatment-related TEAEs.

SECONDARY OUTCOMES:
Dose escalation: maximum tolerated dose (MTD) | Cycle 1 (28 days)
  The MTD will be determined based on safety data.
Maximum plasma concentration (Cmax) | Day 28 for each dose
  Maximum concentration that DT-9081 achieves in plasma
Preliminary anti-tumour activity | From the first dose of study drug until the date of disease progression/recurrence, assessed up to 48 months
  The preliminary anti-tumour activity will be determined based on the assessment of, but not limited to, the objective response rate (ORR). ORR is defined as the percentage of participants with a complete response (CR) or a partial response (PR) at any time during the study according to RECIST v1.1 and immune RECIST (iRECIST).

CONTACTS AND LOCATIONS:
Locations (4):
- Belgium (2):
  - Institut Jules Bordet, Anderlecht
  - Université Catholique de Louvain, Leuven
- France (2):
  - Institut Curie, Paris
  - Institut Claudius Regaud, Toulouse

IPD SHARING:
Plan to Share IPD: No